CLINICAL TRIAL: NCT00271154
Title: REsynchronization reVErses Remodeling in Systolic Left vEntricular Dysfunction (REVERSE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 233
Record Dates: First submitted 2005-12-21; First posted 2005-12-30 (Estimated); Results first posted 2009-05-13 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Implantable Cardioverter Defibrillator; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy; Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT OFF (Placebo Comparator): Cardiac Resynchronization Therapy (CRT) turned OFF in conjunction with optimal medical therapy
  Interventions: Device: Cardiac Resynchronization Therapy (CRT) Device or Implantable Cardioverter Defibrillator (ICD) with CRT
- CRT ON (Active Comparator): Cardiac Resynchronization Therapy (CRT) turned ON in conjunction with optimal medical therapy
  Interventions: Device: Cardiac Resynchronization Therapy (CRT) Device or Implantable Cardioverter Defibrillator (ICD) with CRT

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy (CRT) Device or Implantable Cardioverter Defibrillator (ICD) with CRT — All randomized patients will be implanted with a market-released Medtronic CRT or CRT/ICD device.

SUMMARY:
Heart failure is a progressive disease that decreases the pumping action of the heart. This may cause a backup of fluid in the heart and may result in heart beat changes. When there are changes in the heart beat sometimes an implantable heart device is used to control the rate and rhythm of the heart beat. The purpose of the REVERSE clinical trial is to determine whether pacing in both the left and right ventricles using Cardiac Resynchronization Therapy (CRT) can help slow the progression of heart failure in people who have mild or previous symptoms and poor heart pumping function. This kind of therapy has previously been shown to reduce symptoms and improve exercise capacity in people with more advanced forms of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with previously symptomatic heart failure but no current symptoms (New York Heart Association (NYHA) Class I, Stage C) or subjects with mild heart failure that only sometimes interferes with daily activities (NYHA Class II)
* Subjects with a QRS of 120 ms or more (The QRS interval is a measurement of how the electrical signal involved in a heart beat travels/conducts through the ventricles. A wide QRS (120 ms or more) suggests that there is a conduction problem (or block) in the ventricles).
* Subjects with a left ventricular ejection fraction less than or equal to 40%. (The left ventricular ejection fraction (LVEF) is a measurement of how well the left ventricle pumps blood out to the rest of the body. The higher the LVEF the more blood the ventricle is pumping.)
* Subjects with a left ventricular end diastolic dimension (LVEDD) greater than or equal to 55. (The left ventricular end diastolic dimension (LVEDD) is a measurement of heart size taken during an echocardiogram that is one indication of the health of the left ventricle.)

Exclusion Criteria:

* Subjects who are pacemaker dependent (heart would not beat without the help of an implanted device to pace it).
* Subjects with heart failure that severely limits daily activities (NYHA Class III) or subjects with severe heart failure with symptoms while resting (NYHA Class IV).
* Subjects hospitalized due to heart failure within past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2004-09; Primary Completion 2007-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Linde, MD, PhD, Principal Investigator — Department of Cardiology, Karolinska University Hospital, Stockholm, Sweden
Locations (65):
- United States (34):
  - Huntsville, Alabama
  - Anchorage, Alaska
  - Redwood City, California
  - San Diego, California
  - Atlantis, Florida
  - Jacksonville, Florida
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Ann Arbor, Michigan
  - Saginaw, Michigan
  - Coon Rapids, Minnesota
  - Tupelo, Mississippi
  - Lincoln, Nebraska
  - East Syracuse, New York
  - Manhasset, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Marion, Ohio
  - Doylestown, Pennsylvania
  - Hershey, Pennsylvania
  - West Reading, Pennsylvania
  - Charleston, South Carolina
  - Germantown, Tennessee
  - Kingsport, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Madison, Wisconsin
- Austria (2):
  - Sankt Pölten
  - Weiner Neustadt
- Leuven, Belgium
- Kingston, Ontario, Canada
- Czechia (2):
  - Brno
  - Olomouc
- Denmark (4):
  - Aalborg
  - Aarhus
  - Copenhagen
  - Odense
- France (5):
  - Lyon
  - Marseille
  - Montpellier
  - Nantes
  - Rennes
- Germany (3):
  - Bochum
  - Hamburg
  - Hanover
- Hungary (2):
  - Budapest
  - Szeged
- Dublin, Ireland
- Italy (4):
  - Busto Arsizio
  - Florence
  - Milan
  - Rome
- Kristiansand, Norway
- Spain (2):
  - Madrid
  - Valencia
- Sweden (2):
  - Linköping
  - Stockholm
- Blackpool, United Kingdom

REFERENCES:
- [Result] Linde C, Abraham WT, Gold MR, St John Sutton M, Ghio S, Daubert C; REVERSE (REsynchronization reVErses Remodeling in Systolic left vEntricular dysfunction) Study Group. Randomized trial of cardiac resynchronization in mildly symptomatic heart failure patients and in asymptomatic patients with left ventricular dysfunction and previous heart failure symptoms. J Am Coll Cardiol. 2008 Dec 2;52(23):1834-1843. doi: 10.1016/j.jacc.2008.08.027. Epub 2008 Nov 7. PMID 19038680
- [Result] Linde C, Gold M, Abraham WT, Daubert JC; REVERSE Study Group. Baseline characteristics of patients randomized in The Resynchronization Reverses Remodeling In Systolic Left Ventricular Dysfunction (REVERSE) study. Congest Heart Fail. 2008 Mar-Apr;14(2):66-74. doi: 10.1111/j.1751-7133.2008.07613.x. PMID 18401214
- [Derived] Gold MR, Abraham WT, Butler J, Zile MR, Kahwash R, Gerritse B, Linde C. Win ratio analysis of the REVERSE cardiac resynchronization trial. Heart Rhythm. 2025 Dec;22(12):3042-3049. doi: 10.1016/j.hrthm.2025.04.059. Epub 2025 May 3. PMID 40324513
- [Derived] Fudim M, Dalgaard F, Friedman DJ, Abraham WT, Cleland JGF, Curtis AB, Gold MR, Kutyifa V, Linde C, Ali-Ahmed F, Tang A, Olivas-Martinez A, Inoue LYT, Al-Khatib SM, Sanders GD. Comorbidities and clinical response to cardiac resynchronization therapy: Patient-level meta-analysis from eight clinical trials. Eur J Heart Fail. 2024 Apr;26(4):1039-1046. doi: 10.1002/ejhf.3029. Epub 2023 Sep 15. PMID 37671601
- [Derived] Friedman DJ, Al-Khatib SM, Dalgaard F, Fudim M, Abraham WT, Cleland JGF, Curtis AB, Gold MR, Kutyifa V, Linde C, Tang AS, Ali-Ahmed F, Olivas-Martinez A, Inoue LYT, Sanders GD. Cardiac Resynchronization Therapy Improves Outcomes in Patients With Intraventricular Conduction Delay But Not Right Bundle Branch Block: A Patient-Level Meta-Analysis of Randomized Controlled Trials. Circulation. 2023 Mar 7;147(10):812-823. doi: 10.1161/CIRCULATIONAHA.122.062124. Epub 2023 Jan 26. PMID 36700426
- [Derived] Gold MR, Rickard J, Daubert JC, Cerkvenik J, Linde C. Association of left ventricular remodeling with cardiac resynchronization therapy outcomes. Heart Rhythm. 2023 Feb;20(2):173-180. doi: 10.1016/j.hrthm.2022.11.016. Epub 2022 Nov 25. PMID 36442825
- [Derived] Gold MR, Rickard J, Daubert JC, Zimmerman P, Linde C. Redefining the Classifications of Response to Cardiac Resynchronization Therapy: Results From the REVERSE Study. JACC Clin Electrophysiol. 2021 Jul;7(7):871-880. doi: 10.1016/j.jacep.2020.11.010. Epub 2021 Feb 24. PMID 33640347
- [Derived] Senfield J, Daubert C, Abraham WT, Ghio S, St John Sutton M, Cerkvenik J, Linde C, Gold MR. The Impact of the PR Interval in Patients Receiving Cardiac Resynchronization Therapy: Results From the REVERSE Study. JACC Clin Electrophysiol. 2017 Aug;3(8):818-826. doi: 10.1016/j.jacep.2017.01.017. Epub 2017 Apr 26. PMID 29759777
- [Derived] Linde C, Cleland JGF, Gold MR, Claude Daubert J, Tang ASL, Young JB, Sherfesee L, Abraham WT. The interaction of sex, height, and QRS duration on the effects of cardiac resynchronization therapy on morbidity and mortality: an individual-patient data meta-analysis. Eur J Heart Fail. 2018 Apr;20(4):780-791. doi: 10.1002/ejhf.1133. Epub 2018 Jan 4. PMID 29314424
- [Derived] Gold MR, Padhiar A, Mealing S, Sidhu MK, Tsintzos SI, Abraham WT. Economic Value and Cost-Effectiveness of Cardiac Resynchronization Therapy Among Patients With Mild Heart Failure: Projections From the REVERSE Long-Term Follow-Up. JACC Heart Fail. 2017 Mar;5(3):204-212. doi: 10.1016/j.jchf.2016.10.014. Epub 2017 Jan 11. PMID 28254126
- [Derived] St John Sutton M, Linde C, Gold MR, Abraham WT, Ghio S, Cerkvenik J, Daubert JC; REVERSE Study Group. Left Ventricular Architecture, Long-Term Reverse Remodeling, and Clinical Outcome in Mild Heart Failure With Cardiac Resynchronization: Results From the REVERSE Trial. JACC Heart Fail. 2017 Mar;5(3):169-178. doi: 10.1016/j.jchf.2016.11.012. PMID 28254122
- [Derived] St John Sutton M, Cerkvenik J, Borlaug BA, Daubert C, Gold MR, Ghio S, Chirinos JA, Linde C, Ky B. Effects of Cardiac Resynchronization Therapy on Cardiac Remodeling and Contractile Function: Results From Resynchronization Reverses Remodeling in Systolic Left Ventricular Dysfunction (REVERSE). J Am Heart Assoc. 2015 Sep 11;4(9):e002054. doi: 10.1161/JAHA.115.002054. PMID 26363005
- [Derived] Gold MR, Daubert JC, Abraham WT, Hassager C, Dinerman JL, Hudnall JH, Cerkvenik J, Linde C. Implantable defibrillators improve survival in patients with mildly symptomatic heart failure receiving cardiac resynchronization therapy: analysis of the long-term follow-up of remodeling in systolic left ventricular dysfunction (REVERSE). Circ Arrhythm Electrophysiol. 2013 Dec;6(6):1163-8. doi: 10.1161/CIRCEP.113.000570. Epub 2013 Oct 14. PMID 24125796
- [Derived] Linde C, Daubert C, Abraham WT, St John Sutton M, Ghio S, Hassager C, Herre JM, Bergemann TL, Gold MR; REsynchronization reVErses Remodeling in Systolic left vEntricular dysfunction (REVERSE) Study Group. Impact of ejection fraction on the clinical response to cardiac resynchronization therapy in mild heart failure. Circ Heart Fail. 2013 Nov;6(6):1180-9. doi: 10.1161/CIRCHEARTFAILURE.113.000326. Epub 2013 Sep 6. PMID 24014828
- [Derived] Cleland JG, Abraham WT, Linde C, Gold MR, Young JB, Claude Daubert J, Sherfesee L, Wells GA, Tang AS. An individual patient meta-analysis of five randomized trials assessing the effects of cardiac resynchronization therapy on morbidity and mortality in patients with symptomatic heart failure. Eur Heart J. 2013 Dec;34(46):3547-56. doi: 10.1093/eurheartj/eht290. Epub 2013 Jul 29. PMID 23900696
- [Derived] Linde C, Gold MR, Abraham WT, St John Sutton M, Ghio S, Cerkvenik J, Daubert C; REsynchronization reVErses Remodeling in Systolic left vEntricular dysfunction Study Group. Long-term impact of cardiac resynchronization therapy in mild heart failure: 5-year results from the REsynchronization reVErses Remodeling in Systolic left vEntricular dysfunction (REVERSE) study. Eur Heart J. 2013 Sep;34(33):2592-9. doi: 10.1093/eurheartj/eht160. Epub 2013 May 2. PMID 23641006
- [Derived] Gold MR, Thebault C, Linde C, Abraham WT, Gerritse B, Ghio S, St John Sutton M, Daubert JC. Effect of QRS duration and morphology on cardiac resynchronization therapy outcomes in mild heart failure: results from the Resynchronization Reverses Remodeling in Systolic Left Ventricular Dysfunction (REVERSE) study. Circulation. 2012 Aug 14;126(7):822-9. doi: 10.1161/CIRCULATIONAHA.112.097709. Epub 2012 Jul 10. PMID 22781424
- [Derived] Thebault C, Donal E, Meunier C, Gervais R, Gerritse B, Gold MR, Abraham WT, Linde C, Daubert JC; REVERSE study group. Sites of left and right ventricular lead implantation and response to cardiac resynchronization therapy observations from the REVERSE trial. Eur Heart J. 2012 Nov;33(21):2662-71. doi: 10.1093/eurheartj/ehr505. Epub 2012 Jan 26. PMID 22285578
- [Derived] Gold MR, Linde C, Abraham WT, Gardiwal A, Daubert JC. The impact of cardiac resynchronization therapy on the incidence of ventricular arrhythmias in mild heart failure. Heart Rhythm. 2011 May;8(5):679-84. doi: 10.1016/j.hrthm.2010.12.031. Epub 2010 Dec 23. PMID 21185401
- [Derived] Linde C, Abraham WT, Gold MR, Daubert C; REVERSE Study Group. Cardiac resynchronization therapy in asymptomatic or mildly symptomatic heart failure patients in relation to etiology: results from the REVERSE (REsynchronization reVErses Remodeling in Systolic Left vEntricular Dysfunction) study. J Am Coll Cardiol. 2010 Nov 23;56(22):1826-31. doi: 10.1016/j.jacc.2010.05.055. PMID 21087711
- [Derived] Linde C, Daubert C. Cardiac resynchronization therapy in patients with New York Heart Association class I and II heart failure: an approach to 2010. Circulation. 2010 Sep 7;122(10):1037-43. doi: 10.1161/CIRCULATIONAHA.109.923094. No abstract available. PMID 20823398
- [Derived] St John Sutton M, Ghio S, Plappert T, Tavazzi L, Scelsi L, Daubert C, Abraham WT, Gold MR, Hassager C, Herre JM, Linde C; REsynchronization reVErses Remodeling in Systolic left vEntricular dysfunction (REVERSE) Study Group. Cardiac resynchronization induces major structural and functional reverse remodeling in patients with New York Heart Association class I/II heart failure. Circulation. 2009 Nov 10;120(19):1858-65. doi: 10.1161/CIRCULATIONAHA.108.818724. Epub 2009 Oct 26. PMID 19858419
- [Derived] Daubert C, Gold MR, Abraham WT, Ghio S, Hassager C, Goode G, Szili-Torok T, Linde C; REVERSE Study Group. Prevention of disease progression by cardiac resynchronization therapy in patients with asymptomatic or mildly symptomatic left ventricular dysfunction: insights from the European cohort of the REVERSE (Resynchronization Reverses Remodeling in Systolic Left Ventricular Dysfunction) trial. J Am Coll Cardiol. 2009 Nov 10;54(20):1837-46. doi: 10.1016/j.jacc.2009.08.011. Epub 2009 Oct 1. PMID 19800193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from September 2004 through September 2006 at 73 sites located in the United States, Canada, and Europe.
Pre-assignment Details: A total of 684 patients were enrolled in the study. Of these, 642 patients were attempted for cardiac resynchronization therapy (CRT) device implant. 21 were unsuccessful, leaving 621 patients successfully implanted with a CRT device. Of these 621 patients, 610 were randomized.
Period: Overall Study
Arm/Group | CRT OFF | CRT ON
Started | 191 | 419
Completed | 191 | 419
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRT OFF | CRT ON | Total
Number analyzed (Participants) | 191 | 419 | 610
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 108 | 229 | 337
  >=65 years | 83 | 190 | 273
Age Continuous [Mean (Standard Deviation); unit: years] | 61.8 (11.6) | 62.9 (10.6) | 62.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 92 | 131
  Male | 152 | 327 | 479
Region of Enrollment [Number; unit: participants]
  United States | 108 | 235 | 343
  Spain | 9 | 18 | 27
  Ireland | 1 | 4 | 5
  Austria | 2 | 4 | 6
  United Kingdom | 6 | 9 | 15
  Italy | 5 | 12 | 17
  France | 15 | 34 | 49
  Czech Republic | 0 | 1 | 1
  Hungary | 6 | 13 | 19
  Canada | 1 | 4 | 5
  Belgium | 1 | 3 | 4
  Denmark | 19 | 46 | 65
  Germany | 6 | 11 | 17
  Norway | 3 | 4 | 7
  Sweden | 7 | 17 | 24
  Netherlands | 2 | 4 | 6

OUTCOME MEASURES:

1. Secondary Outcome: Change in Left Ventricular End Systolic Volume, Indexed (LVESVi)
Description: The change is LVESVi measured at 12 months minus LVESVi measured at baseline. The 12-month echocardiographic measurements were made with CRT programmed off, irespective of the treatment assignment. In CRT ON patients these measurements were recorded after a 10 minute washout period. Two core laboratories performed all echo measurements.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: milliliters per meters squared
Arm/Group | CRT OFF | CRT ON
Number analyzed (Participants) | 191 | 419
milliliters per meters squared | -1.3 (23.4) | -18.4 (29.5)
Statistical Analysis 1: Comparison: CRT OFF vs CRT ON; Null hypothesis: mean 12-month change in LVESVi in group 1 = mean 12-month change in LVESVi in group 2; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Primary Outcome: Percentage of Patients Worsened for Clinical Composite Response
Description: Patients considered worsened if they died, were hospitalized with worsening heart failure (HF), crossed over to other arm, demonstrated worsening in New York Heart Association (NYHA) functional class, or reported moderately/markedly worse HF symptoms compared to before CRT implant.
Time Frame: 12 Months
Population: All randomized patients were included using Intent to Treat (ITT).
Measure: Number; unit: Percentage of participants worsened
Arm/Group | CRT OFF | CRT ON
Number analyzed (Participants) | 191 | 419
Percentage of participants worsened | 21.5 | 16
Statistical Analysis 1: Comparison: CRT OFF vs CRT ON; Null hypothesis: Percentage worsened in CRT OFF group = Percentage worsened in CRT ON group; Test type: Superiority or Other; p = 0.10, Chi-squared

ADVERSE EVENTS:
Time Frame: Time of enrollment to 5 years post-implant. All AE's were collected until 12 months (North America) and 24 months (Europe) when only cardiovascular, pulmonary, system, and device-related AE's were collected. AE's reported here are as of 3/5/10.
Description: Serious definition
  * Led to a death,
  * Led to a serious deterioration in health that resulted in:
    * a life-threatening illness or injury,
    * a permanent impairment of a body structure or function
    * hosp. or prolongation of existing hosp.
    * medical or surgical intervention to prevent permanent impairment to body structure or a body function.
Groups:
- Not Randomized: These patients were enrolled in the study, but not randomized to CRT ON or CRT OFF. Their adverse events were collected until they exited the study.
Arm/Group | CRT OFF | CRT ON | Not Randomized
Serious Adverse Events (participants affected / at risk) | 122/191 | 268/419 | 13/38
Other Adverse Events (participants affected / at risk) | 61/119 | 140/491 | 2/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT OFF (N=191) | CRT ON (N=419) | Not Randomized (N=38)
Cardiac failure acute (General disorders) | 30 (52) | 56 (98) | 2 (5)
Medical device change (General disorders) | 19 (19) | 45 (46) | 1 (1)
Ventricular tachycardia (General disorders) | 11 (14) | 30 (43) | 1 (1)
LV lead dislodgement (General disorders) | 13 (15) | 26 (28) | 2 (2)
Chest pain (General disorders) | 4 (4) | 21 (25) | 0 (0)
Pneumonia (General disorders) | 8 (9) | 16 (19) | 1 (1)
Atrial fibrillation (General disorders) | 8 (8) | 15 (19) | 0 (0)
Device lead damage (General disorders) | 8 (8) | 18 (18) | 0 (0)
Inappropriate device therapy (General disorders) | 3 (3) | 16 (16) | 0 (0)
Ventricular fibrillation (General disorders) | 4 (4) | 8 (11) | 1 (1)
Cardiac failure chronic (General disorders) | 5 (6) | 5 (6) | 2 (2)
Chronic obstructive pulmonary disease (General disorders) | 3 (3) | 7 (11) | 0 (0)
RV lead dislodgement (General disorders) | 1 (1) | 13 (13) | 0 (0)
Syncope (General disorders) | 5 (7) | 5 (5) | 1 (1)
Angina pectoris (General disorders) | 4 (4) | 8 (8) | 0 (0)
Atrial flutter (General disorders) | 6 (6) | 4 (5) | 1 (1)
Inappropriate device irritation of tissue (General disorders) | 3 (3) | 9 (9) | 0 (0)
Cerebrovascular accident (General disorders) | 4 (5) | 5 (6) | 0 (0)
Gastrointestinal hemorrhage (General disorders) | 6 (6) | 4 (5) | 0 (0)
Hypotension (General disorders) | 1 (1) | 9 (9) | 1 (1)
Dyspnea (General disorders) | 2 (3) | 7 (7) | 0 (0)
Failure to capture (General disorders) | 5 (6) | 4 (4) | 0 (0)
Lead dislodgement (General disorders) | 0 (0) | 8 (10) | 0 (0)
RA lead dislodgement (General disorders) | 2 (2) | 8 (8) | 0 (0)
Renal failure acute (General disorders) | 4 (4) | 6 (6) | 0 (0)
Transient ischemic attack (General disorders) | 2 (2) | 8 (8) | 0 (0)
Coronary artery disease (General disorders) | 4 (5) | 3 (3) | 0 (0)
Carotid artery stenosis (General disorders) | 2 (2) | 5 (5) | 0 (0)
Implant site hematoma (General disorders) | 1 (1) | 6 (6) | 0 (0)
Myocardial infarction (General disorders) | 3 (3) | 4 (4) | 0 (0)
Osteoarthritis (General disorders) | 2 (2) | 5 (5) | 0 (0)
Pneumothorax (General disorders) | 0 (0) | 5 (6) | 0 (0)
Acute myocardial infarction (General disorders) | 1 (1) | 4 (4) | 0 (0)
Atrial tachycardia (General disorders) | 1 (1) | 3 (3) | 1 (1)
Ischemic stroke (General disorders) | 0 (0) | 3 (5) | 0 (0)
Pericardial effusion (General disorders) | 2 (2) | 3 (3) | 0 (0)
Peripheral vascular disorder (General disorders) | 1 (3) | 1 (1) | 1 (1)
Renal failure (General disorders) | 2 (2) | 3 (3) | 0 (0)
Sudden cardiac death (General disorders) | 2 (2) | 3 (3) | 0 (0)
Acute pulmonary edema (General disorders) | 0 (0) | 3 (3) | 1 (1)
Anemia (General disorders) | 0 (0) | 4 (4) | 0 (0)
Asthma (General disorders) | 0 (0) | 2 (3) | 1 (1)
Atrioventricular block complete (General disorders) | 0 (0) | 1 (1) | 3 (3)
Bradycardia (General disorders) | 1 (1) | 3 (3) | 0 (0)
Bronchitis (General disorders) | 0 (0) | 3 (4) | 0 (0)
Cardiac arrest (General disorders) | 2 (2) | 2 (2) | 0 (0)
Cholecystitis acute (General disorders) | 2 (2) | 2 (2) | 0 (0)
Deep vein thrombosis (General disorders) | 2 (2) | 2 (2) | 0 (0)
Implant site infection (General disorders) | 2 (2) | 1 (2) | 0 (0)
Inappropriate device signal detection (General disorders) | 3 (3) | 1 (1) | 0 (0)
Ischemic cardiomyopathy (General disorders) | 1 (1) | 2 (2) | 1 (1)
Lung neoplasm malignant (General disorders) | 2 (2) | 2 (2) | 0 (0)
Respiratory failure (General disorders) | 1 (1) | 3 (3) | 0 (0)
Acute respiratory failure (General disorders) | 2 (2) | 1 (1) | 0 (0)
Angina unstable (General disorders) | 0 (0) | 3 (3) | 0 (0)
Aortic aneurysm (General disorders) | 2 (2) | 1 (1) | 0 (0)
Atrioventricular block third degree (General disorders) | 1 (1) | 2 (2) | 0 (0)
Back pain (General disorders) | 1 (1) | 2 (2) | 0 (0)
Bronchitis acute (General disorders) | 0 (0) | 3 (3) | 0 (0)
Cardiac perforation (General disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiac tamponade (General disorders) | 1 (1) | 1 (1) | 1 (1)
Contusion (General disorders) | 1 (1) | 1 (1) | 1 (1)
Defibrillation threshold increased (General disorders) | 1 (1) | 2 (2) | 0 (0)
Dehydration (General disorders) | 1 (1) | 2 (2) | 0 (0)
Dizziness (General disorders) | 0 (0) | 2 (3) | 0 (0)
Esophageal carcinoma (General disorders) | 0 (0) | 3 (3) | 0 (0)
Hematoma (General disorders) | 0 (0) | 3 (3) | 0 (0)
Intracardiac thrombus (General disorders) | 1 (1) | 2 (2) | 0 (0)
Myocardial ischemia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3) | 0 (0)
Pericarditis (General disorders) | 0 (0) | 2 (3) | 0 (0)
Presyncope (General disorders) | 1 (1) | 2 (2) | 0 (0)
Prostate examination abnormal (General disorders) | 0 (0) | 3 (3) | 0 (0)
Pulmonary edema (General disorders) | 2 (2) | 1 (1) | 0 (0)
Subclavian vein thrombosis (General disorders) | 1 (1) | 2 (2) | 0 (0)
Therapeutic agent toxicity (General disorders) | 1 (2) | 1 (1) | 0 (0)
Anxiety (General disorders) | 0 (0) | 1 (1) | 1 (1)
Aortic stenosis (General disorders) | 1 (1) | 1 (1) | 0 (0)
Arrhythmia supraventricular (General disorders) | 0 (0) | 2 (2) | 0 (0)
Arteriovenous fistula (General disorders) | 0 (0) | 1 (1) | 1 (1)
Biliary colic (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (General disorders) | 0 (0) | 2 (2) | 0 (0)
Coronary artery dissection (General disorders) | 0 (0) | 2 (2) | 0 (0)
Coronary artery stenosis (General disorders) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus (General disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (General disorders) | 1 (1) | 1 (1) | 0 (0)
Drug hypersensitivity (General disorders) | 1 (1) | 1 (1) | 0 (0)
Drug toxicity (General disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspnea exertional (General disorders) | 1 (1) | 1 (1) | 0 (0)
Electromechanical dissociation (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
Heart transplant (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycemia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Inappropriate device stimulation of tissue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Mental status changes (General disorders) | 1 (1) | 1 (1) | 0 (0)
Mitral valve incompetence (General disorders) | 0 (0) | 1 (2) | 0 (0)
Orthostatic hypotension (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oversensing (General disorders) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia aspiration (General disorders) | 0 (0) | 2 (2) | 0 (0)
Postoperative wound infection (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (General disorders) | 0 (0) | 1 (2) | 0 (0)
Pulmonary fibrosis (General disorders) | 0 (0) | 1 (2) | 0 (0)
Sepsis (General disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope vasovagal (General disorders) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (General disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal abscess (General disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety disorder (General disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial disorder (General disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial stenosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriogram coronary (General disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriopathic disease (General disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Biopsy liver (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac ablation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac procedure complication (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-renal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy alcoholic (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical dysplasia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (General disorders) | 1 (1) | 0 (0) | 0 (0)
Colonic obstruction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Colostomy (General disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Contrast media reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery restenosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased RV Sensing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Device electrical finding (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device migration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device related infection (General disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus insulin-dependent (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dislodgement of LV lead (General disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis esophageal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Elevated pacing threshold (General disorders) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Goiter (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hairy cell leukemia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma evacuation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hemianopsia homonymous (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypervolemic (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site erosion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0)
In-stent arterial restenosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Incision site complication (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia repair (General disorders) | 0 (0) | 1 (1) | 0 (0)
Intermittent claudication (General disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Iodine allergy (General disorders) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (General disorders) | 1 (1) | 0 (0) | 0 (0)
Leukothrombopenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Low cardiac output syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection viral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lung consolidation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (General disorders) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (General disorders) | 0 (0) | 1 (1) | 0 (0)
Metastatic neoplasm (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve disease (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve repair (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasm malignant (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nodal arrhythmia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (General disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (General disorders) | 0 (0) | 1 (1) | 0 (0)
Perianal abscess (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischemia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pituitary tumor (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (General disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (General disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Renal cancer metastatic (General disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (General disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (General disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal hemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (General disorders) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer stage unspecified (General disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Spondylolysis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid hemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Subdural hematoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Throat lesion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillar disorder (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth disorder (General disorders) | 0 (0) | 1 (1) | 0 (0)
Twiddler's syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary bladder adenoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Valvuloplasty cardiac (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (General disorders) | 0 (0) | 1 (1) | 0 (0)
Venous stenosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular assist device insertion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo CNS origin (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vestibular neuronitis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Viral infection (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord polyp (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vocal cord thickening (General disorders) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT OFF (N=119) | CRT ON (N=491) | Not Randomized (N=38)
Cardiac failure chronic (General disorders) | 24 (30) | 31 (35) | 1 (1)
Atrial fibrillation (General disorders) | 8 (8) | 47 (57) | 0 (0)
Dizziness (General disorders) | 9 (9) | 25 (29) | 1 (1)
Inappropriate device stimulation of tissue (General disorders) | 11 (12) | 21 (25) | 0 (0)
Inappropriate device irritation of tissue (General disorders) | 4 (4) | 26 (30) | 1 (1)
Hypotension (General disorders) | 10 (12) | 16 (16) | 0 (0)
Fatigue (General disorders) | 12 (12) | 15 (15) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators to publish study results per the publication plan/protocol following Medtronic's review to determine whether confidential information ("CI") is disclosed. Any such CI is deleted prior to publication/presentation. Medtronic may not censor/interfere with the publication except as described. Investigators may not publish any single-site publications until the main multi-site study publication has occurred.